CLINICAL TRIAL: NCT05154968
Title: A Study to Evaluate Injection-Site Pain of Two Formulations (Both Refrigerated and Room Temperature) Using an Autoinjector Device in Healthy Subjects
Brief Title: A Study of Two Formulations (Both Refrigerated and Room Temperature) Using an Autoinjector Device in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 18167; J3G-MC-S003 (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-11-19; First posted 2021-12-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Sodium Chloride; Mannitol

STUDY DESIGN:
Who Masked: Participant
Masking Description: Partially blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (ABCD) (Experimental): Participants will receive 1 millilitre (ml) subcutaneous (SC) injection of treatment A (higher pain refrigerated solution is a formulation matrix solution of an acidic solution citrate buffer and sodium chloride at the potential of hydrogen (pH) 5.7) followed by treatments B (higher pain Room Temperature [RT] solution is a formulation matrix solution of an acidic solution containing citrate buffer and sodium chloride at pH 5.7), C (lower pain refrigerated solution contains mannitol), and D (lower pain RT solution contains mannitol) in the right upper quadrant, left upper quadrant, right lower quadrant, and left lower quadrant respectively using a prefilled autoinjector device.
  Interventions: Drug: Sodium chloride; Drug: Citrate buffer; Drug: Mannitol; Device: Prefilled Autoinjector
- Sequence 2 (BDAC) (Experimental): Participants will receive 1 ml SC injection of treatment B (higher pain RT solution is a formulation matrix solution of an acidic solution containing citrate buffer and sodium chloride at pH 5.7) followed by treatments D (lower pain RT solution contains mannitol), A (higher pain refrigerated solution is a formulation matrix solution of an acidic solution citrate buffer and sodium chloride at pH 5.7), and C (lower pain refrigerated solution contains mannitol) in the right upper quadrant, left upper quadrant, right lower quadrant, and left lower quadrant respectively using a prefilled autoinjector device.
  Interventions: Drug: Sodium chloride; Drug: Citrate buffer; Drug: Mannitol; Device: Prefilled Autoinjector
- Sequence 3 (CADB) (Experimental): Participants will receive 1 ml SC injection of treatment C (lower pain refrigerated solution contains mannitol) followed by treatments A (higher pain refrigerated solution is a formulation matrix solution of an acidic solution citrate buffer and sodium chloride at pH 5.7), D (lower pain RT solution contains mannitol), and B (higher pain RT solution is a formulation matrix solution of an acidic solution containing citrate buffer and sodium chloride at pH 5.7) in the right upper quadrant, left upper quadrant, right lower quadrant, and left lower quadrant respectively using a prefilled autoinjector device.
  Interventions: Drug: Sodium chloride; Drug: Citrate buffer; Drug: Mannitol; Device: Prefilled Autoinjector
- Sequence 4 (DCBA) (Experimental): Participants will receive 1 ml SC injection of treatment D (lower pain RT solution contains mannitol) followed by treatments C (lower pain refrigerated solution contains mannitol), B (higher pain RT solution is a formulation matrix solution of an acidic solution containing citrate buffer and sodium chloride at pH 5.7), and A (higher pain refrigerated solution is a formulation matrix solution of an acidic solution citrate buffer and sodium chloride at pH 5.7), in the right upper quadrant, left upper quadrant, right lower quadrant, and left lower quadrant respectively using a prefilled autoinjector device.
  Interventions: Drug: Sodium chloride; Drug: Citrate buffer; Drug: Mannitol; Device: Prefilled Autoinjector

INTERVENTIONS:
Drug: Sodium chloride — Administered SC infusion.
Drug: Citrate buffer — Administered SC infusion.
Drug: Mannitol — Administered SC infusion.
Device: Prefilled Autoinjector — Used to administer the drug through SC infusion.

SUMMARY:
The main purpose of the study is to assess the injection site pain intensity of two formulations using prefilled autoinjector device in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker
* BMI greater than (>)18.5 and less than (<) 30.0 kilograms per square meter (kg/m2)
* Body weight greater than or equal to (≥) 50.0 kg for males and ≥45.0 kg for females
* Are in good health, as determined by the investigator (or designee) to have no clinically significant findings from medical and surgical history, physical examination, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations
* Are reliable and willing to make themselves available for the duration of the study, are willing to follow study procedures, and demonstrate the ability to self-inject

Exclusion Criteria:

* Are pregnant or breastfeeding
* Have a positive urine drug screen or alcohol breath test at screening Have participated in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing or concomitant participation in an investigational study involving no drug or device administration
* Have known allergic reactions to any components of mannitol or the placebo matrix or related compounds or history of significant atopy
* Have self-perceived dullness or loss of sensation on either side of the body or the abdomen
* Have tattoos or scars over the abdomen or other factors (e.g., rash, excessive folds of skin) that, in the Investigator's opinion, would interfere with injection site assessments
* Are currently using painkillers, aspirin, or other non-steroidal anti-inflammatory drugs (NSAIDs). Intend to use prescription or over-the-counter medication for pain or inflammation within 7 days prior to the first injection
* Have any reason which, in the opinion of the Investigator, would prevent the participant from participating in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) Pain score at Injection Site at Time Zero (T0) | within 1 minute post injection
  The Infusion site pain VAS score is a participant administered single item scale designed to measure pain using a 0-100 millimeter (mm) horizontal VAS. Overall severity of participant's pain is indicated by placing a single mark on the horizontal 100 mm scale from 0 mm (no pain) to 100 mm (worst possible pain).

SECONDARY OUTCOMES:
Visual analogue scale (VAS) Pain score at Injection Site after Time Zero (T0) | within 5, 10, 15, 30 and 60 minutes post injection
  The Infusion site pain VAS score is a participant administered single item scale designed to measure pain using a 0-100 millimeter (mm) horizontal VAS. Overall severity of participant's pain is indicated by placing a single mark on the horizontal 100 mm scale from 0 mm (no pain) to 100 mm (worst possible pain).
Number of Participants with Injection Site Reactions (ISR) | 10 and 60 minutes post injection
  ISR will consists of rating the severity of skin reaction at the injection site using the scores below 0=no reaction, 1= easily tolerated erythema and/or light bruising, 2= distributing erythema with swelling and/or distributing bruising, 3=almost intolerable symptoms, or clinically definite skin necrosis, characterized by any of the following: oozing, weeping, skin breakdown, ulceration, scar formation. Higher the score worst the injection site reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Eli Lilly and Company
Locations (1):
- Syneos Health, Québec, Canada

IPD SHARING:
Plan to Share IPD: No